CLINICAL TRIAL: NCT04603092
Title: Digital Health Literacy Intervention by Community Health Workers for Corona Preventive Behaviors for Disadvantaged Women at Primary Level
Brief Title: Digital Health Literacy Intervention for Disadvantaged Women During Corona
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Forman Christian College, Pakistan (Other)
Collaborators: doctHERs (Industry); Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Sara Rizvi Jafree, Assistant Professor, Department of Sociology, Forman Christian College, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FormanChristianC
Record Dates: First submitted 2020-10-19; First posted 2020-10-26 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Health Literacy
Keywords: digital health literacy; community healthcare workers; coronavirus; primary healthcare; maternal and child health
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: The control and experiment group will both be provided a hard-copy of a health literacy booklet and electronically administered the: (a) base-line survey, and (b) the pre-test survey and the post-test survey.
  The experiment group will receive a digital health literacy intervention in two target areas: (i) hygiene and sanitation, and (ii) coronavirus awareness and prevention.
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Disadvantaged women in primary setting receiving digital health literacy intervention (Experimental): The study population will comprise of disadvantaged women dependent on primary healthcare services, who do not have access to digital tools (smartphone, computer, laptop) or Wifi in their home. This group will receive the digital health literacy intervention.
  Interventions: Behavioral: Digital Health Literacy Intervention
- Disadvantaged women in primary setting not receiving digital health literacy intervention (No Intervention): The study population will comprise of disadvantaged women dependent on primary healthcare services, who do not have access to digital tools (smartphone, computer, laptop) or Wifi in their home. This control group will not receive the digital health literacy intervention.

INTERVENTIONS:
Behavioral: Digital Health Literacy Intervention — Willing women participants will be provided equipment with instructions for the intervention, including a smartphone and a 4G Wifi gadget. The health literacy intervention, delivered to the experiment group, will last three months and will include a combination of the following four components:
  Component 1: Health literacy video tutorial. Component 2: Virtual one-on-one weekly meetings. Component 3: Monthly group virtual meetings and Whatsapp group. Component 4: Provision and guidance of a self-management chart.
  Arms: Disadvantaged women in primary setting receiving digital health literacy intervention

SUMMARY:
The aim is to deliver a digital health literacy intervention to disadvantaged women to improve their health behaviors with regard to (i) hygiene and sanitation, and (ii) coronavirus awareness and prevention in four provinces of Pakistan through women community health workers.

DETAILED DESCRIPTION:
There is a need to continue primary healthcare services through digital communication for disadvantaged women living in underdeveloped areas of Pakistan, especially in the age of coronavirus pandemic, social distancing, and lockdown of communities. This project will be the first of its kind in aiming to provide women with a smartphone and digital access for a digital health literacy intervention through community healthcare workers. The majority of poor women in Pakistan who are dependent on primary health services: 1. suffer from health challenges more than men due to multiple social and structural disadvantages, 2. are the dominant care-providers and nurturers in the home, and 3. need support in understanding public health messages during health crises due to low health literacy and awareness. The digital health literacy intervention will be delivered in target two areas: (i) hygiene and sanitation, and (ii) coronavirus awareness and prevention. Women will be sampled from disadvantaged areas across the four provinces of Pakistan- Baluchistan, KPK, Punjab, and Sindh. A target of 1,000 women will comprise the sample with 500 women each assigned to the control and experiment group.

ELIGIBILITY:
Inclusion Criteria:

* Disadvantaged women dependent on primary healthcare services
* Women of the reproductive age group, 15 years to 49 years

Exclusion Criteria:

* Women above 49 years

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1010 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Changes in health directed behavior | 3 months
  A total of 135 questions will be used, with five domains being covered through the following surveys: (i) Health Education Impact Questionnaire, (ii) Survey on Hygiene Knowledge, Attitude and Practice, (iii) Homecare of Covid Survey, (iv) Survey for mobile u-Health program by Ahn, Bae, and Kim and (v) Women's Health Care Experiences Survey. It is a five-point Likert-type scale (strongly agree - agree - neutral - disagree - strongly disagree). The highest value of the scale is 6 and the lowest value is 1; with 6 points showing strong agreement with the item statement (E.g. Q80. We are cleaning the eating, drinking, and cooking utensil with dish detergent after every use).

CONTACTS AND LOCATIONS:
Locations (1):
- Forman Christian College University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The SPSS data set will be publicly available. No names of participants will be taken during data collection. Participants will be allocated a code.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months

REFERENCES:
- [Derived] Jafree SR, Bukhari N, Muzamill A, Tasneem F, Fischer F. Digital health literacy intervention to support maternal, child and family health in primary healthcare settings of Pakistan during the age of coronavirus: study protocol for a randomised controlled trial. BMJ Open. 2021 Mar 2;11(3):e045163. doi: 10.1136/bmjopen-2020-045163. PMID 33653760